CLINICAL TRIAL: NCT00909090
Title: Effects of Lutein and Zeaxanthin Upon MPOD and Its Effects Upon Glare Disability, Photostress Recovery, and Contrast Enhancement in Healthy Subjects: A Randomized, Double-blind Placebo-controlled Study
Brief Title: Macular Pigment and Glare Disability
Acronym: MP-GD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Billy R. Hammond, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UGA-2009-10141-1
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Vision, Entoptic
Keywords: macular pigment; glare disability; lutein; photostress; chromatic contrast sensitivity
MeSH Terms: interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Intervention Model Description: Two arms: nutritional supplement vs. placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin
  Interventions: Dietary Supplement: 12 mg Lutein + Zeaxanthin
- Placebo (Placebo Comparator): visually identical placebo
  Interventions: Dietary Supplement: Visually identical placebo

INTERVENTIONS:
Dietary Supplement: 12 mg Lutein + Zeaxanthin — 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin, taken once daily for one year
  Other Names: FloraGlo lutein + OptiSharp zeaxanthin
  Arms: Intervention
Dietary Supplement: Visually identical placebo — Visually identical placebo, taken once daily for one year
  Arms: Placebo

SUMMARY:
The purpose of this study is:

I. To measure MP optical density (MPOD) in two groups (experimental and placebo) of 50 subjects each (N = 100), during an Lutein + Zeaxanthin supplementation period of 12 months.

II. To test the hypothesis that increases in MP (via 12 mg daily Lutein + Zeaxanthin supplementation) will result in significantly improved visual performance under disability glare conditions.

III. To test the hypothesis that increases in MP (via 12 mg daily L + Z supplementation) will result in significantly reduced photostress recovery times.

IV. To test the hypothesis that increases in MP (via 12 mg daily L + Z supplementation) will result in improved contrast enhancement.

DETAILED DESCRIPTION:
The following measurements will be taken, before and after supplementation with lutein and zeaxanthin:

Macular pigment optical density (MPOD) Visual performance under glare conditions Photostress recovery times chromatic contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Age: 18 - 40 years
* BMI: 20-30
* No anticipated changes in dieting habits (as relevant to xanthophyll intake).
* No anticipated surgical procedures.
* Assessed as healthy, based on a pre-study examination including medical history, physical examination, and clinical laboratory. The examination will be performed by an MD or a Nurse Practitioner.
* Willingness and ability to give written informed consent and willingness and ability to comply with the study requirements.
* Corrected visual acuity (ETDRS): better than 20/60

Exclusion Criteria:

* BMI <20 or >30
* Age <18 or >40 years
* Smokers
* Current or history of relevant diseases (such as AMD)
* Corrected visual acuity worse than 20/60
* Inability to reliably perform MPOD measurements by heterochromatic flicker photometry or any of the other ophthalmic tests of the study.
* Any condition likely to interfere with normal gastro-intestinal absorption of xanthophylls.
* Current use of xanthophyll containing supplements
* Use of xanthophyll containing supplements in the past 6 months
* Participation in any other study during last 1 month.
* Blood donation during the last 3 months.
* Known hypersensitivity or allergy to xanthophylls.
* Regular intake of medications or supplements, which the principal investigator deems likely to confound the study outcomes.
* Suspected lack of compliance with any requirements of the study.
* Childbearing potential and unwillingness to refrain from acceptable anticonceptive measures (not including abstinence).
* Current pregnancy or breast feeding
* Any relevant abnormalities in the routine laboratory tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male, female, other, non-conforming
Enrollment: 109 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Billy R Hammond, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- Vision Sciences Laboratory, UGA, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammond BR, Fletcher LM, Roos F, Wittwer J, Schalch W. A double-blind, placebo-controlled study on the effects of lutein and zeaxanthin on photostress recovery, glare disability, and chromatic contrast. Invest Ophthalmol Vis Sci. 2014 Dec 2;55(12):8583-9. doi: 10.1167/iovs.14-15573. PMID 25468896
- [Derived] Hammond BR Jr, Fletcher LM, Elliott JG. Glare disability, photostress recovery, and chromatic contrast: relation to macular pigment and serum lutein and zeaxanthin. Invest Ophthalmol Vis Sci. 2013 Jan 17;54(1):476-81. doi: 10.1167/iovs.12-10411. PMID 23211814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated in May, 2009. The enrollment period was rolling and lasted for 30 months. Enrollment closed in November, 2011. Participants were recruited from the local Athens, Clarke-County community and the University of Georgia student population.
Pre-assignment Details: Key events:
  Telephone screening to confirm eligibility Enrollment Randomization
Groups:
- Intervention: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin
  Intervention: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin, taken once daily for one year
- Placebo: visually identical placebo
  Placebo: Visually identical placebo, taken once daily for one year
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 53 | 56
Completed | 36 | 39
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- 12 mg Lutein + Zeaxanthin: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin
  Intervention: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin, taken once daily for one year
- Visually Identical Placebo: visually identical placebo
  Placebo: Visually identical placebo, taken once daily for one year
- Total: Total of all reporting groups
Arm/Group | 12 mg Lutein + Zeaxanthin | Visually Identical Placebo | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (4.61) | 22.7 (3.32) | 23.2 (3.97)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 22 | 22 | 44
  Gender: Female | 31 | 34 | 65
Region of Enrollment [Number; unit: participants]
  United States | 53 | 56 | 109
BMI [Mean (Standard Deviation); unit: kg/cm^2] — Body mass index, computed from height (cm) and weight (kg)
  kg/cm^2 | 22.9 (2.45) | 22.8 (2.66) | 22.85 (2.56)
Iris Darkness [Mean (Standard Deviation); unit: units on a scale] — Visual inspection of iris color and comparison to an iris color scale on a computer monitor. Darkest irides score 1-2; Lightest irides score 4-5.
  units on a scale | 2.90 (1.31) | 2.81 (1.27) | 2.86 (1.29)

OUTCOME MEASURES:

1. Primary Outcome: Macular Pigment Optical Density
Description: optical density of macular pigment layer of the neural retina at 30-minutes of retinal eccentricity
Time Frame: every three months for one year; 12-month measure reported.
Population: Participants who completed all four measurements
Measure: Mean (Standard Deviation); unit: optical density
Groups:
- Luten + Zeaxanthin: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin
  Intervention: 10 mg FloraGlo lutein + 2 mg Optisharp zeaxanthin, taken once daily for one year
Arm/Group | Luten + Zeaxanthin | Placebo
Number analyzed (Participants) | 36 | 39
optical density | 0.54 (0.10) | 0.42 (0.10)
Statistical Analysis 1: Comparison: Luten + Zeaxanthin vs Placebo; Test type: Superiority; p = 0.01, t-test, 2 sided

2. Secondary Outcome: Glare Disability
Description: light energy needed to obscure or veil a visual target; calculated as log-relative energy, which is the physical energy needed for the subject to report that the visual target has been veiled, given the intensity of the target, logged.
Time Frame: 12-month data point only
Measure: Mean (Standard Deviation); unit: log relative energy
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 36 | 39
log relative energy | 1.81 (0.10) | 1.83 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Analysis compared mean differences between placebo and intervention at the 12-month time point; Test type: Superiority; p = 0.21, Regression, Linear

3. Secondary Outcome: Photostress Recovery Time
Description: amount of time needed to recover from exposure to a bright light, and to regain sight of a visual target
Time Frame: improvement in recovery time; baseline recovery time (sec) minus 12-month recovery time (sec)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 12 mg Lutein + Zeaxanthin | Visually Identical Placebo
Number analyzed (Participants) | 36 | 39
seconds | 10.5 (7.5) | 4.5 (6.0)
Statistical Analysis 1: Comparison: 12 mg Lutein + Zeaxanthin vs Visually Identical Placebo; Analysis compared mean change from baseline to 12-month time points; Test type: Superiority; p = 0.01, t-test, 1 sided

4. Secondary Outcome: Heterochromatic Contrast Sensitivity
Description: amount of short-wave light energy necessary to obscure of veil a visual target, calculated as log-relative energy, which is the physical energy needed for the subject to report that the visual target has been veiled, given the intensity of the target, logged.
Time Frame: 12-month data point only
Measure: Mean (Standard Deviation); unit: log relative energy
Arm/Group | 12 mg Lutein + Zeaxanthin | Visually Identical Placebo
Number analyzed (Participants) | 36 | 39
log relative energy | 1.21 (0.14) | 1.16 (0.10)
Statistical Analysis 1: Comparison: 12 mg Lutein + Zeaxanthin vs Visually Identical Placebo; analysis conducted on mean change over one year, between groups; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: One year
Description: Adverse event collection occurred over the phone at one month intervals, and during in-person follow-up visits every three months.
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/56
Other Adverse Events (participants affected / at risk) | 0/53 | 0/56

LIMITATIONS AND CAVEATS:
Sample included only young, healthy adults with acute vision. Because the sample was recruited from the local college student population, there were high rates of attrition (students moving away, forgetting appointments, discontinuing contact)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No